CLINICAL TRIAL: NCT05309369
Title: Musical Engagement of Brain LObes in Alzheimer's Disease Patients StudY
Acronym: MELODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency); American Association of Retired Persons (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00115303
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Dementia; Music Therapy
Keywords: Dementia; Alzheimer Disease; Brain stimulation; Music
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred Music - Visit 1, Nature Sounds - Visit 2 (Experimental)
  Interventions: Behavioral: Preferred Music; Behavioral: Nature Sounds
- Nature Sounds - Visit 1, Preferred Music - Visit 2 (Placebo Comparator)
  Interventions: Behavioral: Preferred Music; Behavioral: Nature Sounds

INTERVENTIONS:
Behavioral: Preferred Music — Participants will listen to selected music using over-ear headphones delivered as 10-minute segments at the top of each hour over the course of 3 hours
Behavioral: Nature Sounds — Participants will listen to nature sounds using over-ear headphones delivered as 10-minute segments at the top of each hour over the course of 3 hours

SUMMARY:
This is a randomized, cross-over study to measure global and clinical impact and level of arousal in subjects suffering from moderate to severe Alzheimer's disease when exposed to emotionally impactful music compared to control intervention.

DETAILED DESCRIPTION:
In partnership with the study partner (a person who spends 10 hours or more a week with the subject and can reliably report on the subject's condition), three tunes will be chosen for the purposes of the study. The tunes chosen will need to be related to a past meaningful, positive experience of the subject, as determined by the subject and the subject's study partner. The pieces will be restricted in duration to between 1.5 and 2 minutes each. A piece will be chosen at random and will be saved on a portable device, and subjects will be asked to listen to the melody using high quality, over-ear headphones. The total exposure time will be 10 minutes each hour over a three-hour period. The melody will be repeated as many times as necessary to complete the 10-minute period. The control intervention will involve listening to nature sounds at the same duration and administration scheme. Functional magnetic resonance imaging will be used to identify how brain networks are modulated via exposure to this music and how they associate with the clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Person of any sex/gender aged between 55 and 90
* Stated willingness to comply with all study procedures and availability for the duration of the study
* In the opinion of the investigator, has an informant able and willing to provide accurate information about the participant (may be paid or unpaid caregiver)
* Suffer from moderate to severe Alzheimer's disease as established by the study team using the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) Alzheimer's Criteria for possible and probable Alzheimer's Disease
* Diagnosis of Alzheimer's disease or other type of dementia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
* Mini Mental State Examination (MMSE) score of 5-20
* Subject is reported by the study partner to be able to listen to a minimum of 10 minutes of music and a sound in an uninterrupted manner.

Exclusion Criteria:

* Suffer from severe hearing impairment as reported by the informant
* Presence of neuropsychiatric symptoms of dementia as determined by clinical observation by the Principal Investigator, including history of agitation and/or combative behavior.
* Individuals who score ≥ 12 seconds on the Timed Up and Go (TUG) Test.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Mintzer, MD, MBA, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will be part of the Alzheimer's Clinical Trials Consortium (ACTC). The study abides by the principles for sharing of research data as described in the NIH Public Access Policy on data sharing. The researchers endorse the sharing of final de-identified research data to serve important scientific goals. This project will facilitate sharing of software, archived study datasets (including images), assessment instruments, forms, and procedures through the web-based tools of the ACTC. The ACTC web portal will include access to inventories of resources and request procedures. All ACTC archival datasets will be included on the Global Alzheimer's Association Interactive Network (GAAIN); ACTC data can be accessed via the GAAIN platform; full or partial archived datasets can be shared via the dedicated ACTC Dataset- Sharing Portal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It will become available one year after study recruitment it completed.

REFERENCES:
- [Derived] Mintzer J, Long R, Fritts A, Joseph J, Nietert PJ, Calev N, Brawman-Mintzer O. Musical Engagement of brain LObes in Alzheimer's Disease patients study (MELODY): A randomized controlled trial. Int Psychogeriatr. 2025 Dec;37(6):100087. doi: 10.1016/j.inpsyc.2025.100087. Epub 2025 May 24. PMID 40414740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI contacted physicians in the Charleston, South Carolina area to inform them about the study and request patient referrals of potential participants. Once a referral was made, the potential participant was contacted by the PI via telephone, the study was described, and if the participant and study partner expressed interest in the study, the study coordinator scheduled them for a Screening Visit.
Pre-assignment Details: No significant events in the study occured after participant enrollment and prior to assignment of participants to an arm or group.
Period: First Intervention (1 Week)
Arm/Group | Preferred Music - Visit 1, Nature Sounds - Visit 2 | Nature Sounds - Visit 1, Preferred Music - Visit 2
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Preferred Music - Visit 1, Nature Sounds - Visit 2 | Nature Sounds - Visit 1, Preferred Music - Visit 2
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preferred Music - Visit 1, Nature Sounds - Visit 2 | Nature Sounds - Visit 1, Preferred Music - Visit 2 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Intervention Response as Evaluated by the Clinical Global Impression of Change (CGIC)
Description: This is a 7-item score ranging from "markedly worse" to "markedly improved". It is assessed by the study clinician who interviews both participant and makes an informed judgment how to incorporate their input.
Time Frame: Visit 1 (Day 14 +/- 3 days), Visit 2 (Day 21 +/- 3 days)
Population: All 10 participants were assessed after being exposed to preferred music (PM) and nature sounds (NS) and rated on the Clinical Global Impression of Change (CGIC).
Measure: Count of Participants; unit: Participants
Arm/Group | Preferred Music | Nature Sounds
Number analyzed (Participants) | 10 | 10
Participants
  Marked improvement - Rating 1 | 0 | 0
  Moderate improvement - Rating 1 | 5 | 2
  Minimal improvement - Rating 1 | 2 | 0
  No change - Rating 1 | 1 | 4
  Minimal worsening - Rating 1 | 1 | 1
  Moderate worsening - Rating 1 | 1 | 3
  Marked worsening - Rating 1 | 0 | 0
  Marked improvement - Rating 2 | 0 | 0
  Moderate improvement - Rating 2 | 9 | 2
  Minimal Improvement - Rating 2 | 1 | 0
  No Change - Rating 2 | 0 | 2
  Minimal worsening - Rating 2 | 0 | 2
  Moderate worsening - Rating 2 | 0 | 4
  Marked worsening - Rating 2 | 0 | 0

2. Secondary Outcome: Change in Level of Arousal as Evaluated by the Stanford Sleepiness Scale (SSS)
Description: Participants will provide a self-assessed scoring of their level of arousal on a scale of 1-7 ranging from "Feeling active, vital, alert, or wide awake" to "No longer fighting sleep, sleep onset soon; having dream-like thoughts".
Time Frame: Visit 1 (Day 14 +/- 3 days), Visit 2 (Day 21 +/- 3 days)
Population: All 10 participants were assessed after being exposed to preferred music (PM) and nature sounds (NS) and rated on the Stanford Sleepiness Scale (SSS).
Measure: Count of Participants; unit: Participants
Arm/Group | Preferred Music | Nature Sounds
Number analyzed (Participants) | 10 | 10
Participants
  1 - Feeling active, vital, alert, or wide awake - Rating 1 | 3 | 1
  2 - Functioning at high levels, but not at peak - Rating 1 | 1 | 4
  3 - Awake, but relaxed; responsive, but not fully alert - Rating 1 | 5 | 2
  4 - Somewhat foggy, let down - Rating 1 | 0 | 2
  5 - Foggy; losing interest in staying awake; slowed down - Rating 1 | 1 | 1
  6 - Sleepy, woozy, fighting sleep; prefer to lie down - Rating 1 | 0 | 0
  7 - No longer fighting sleep; sleep onset soon - Rating 1 | 0 | 0
  X - Asleep - Rating 1 | 0 | 0
  1 - Feeling active, vital, alert, or wide awake - Rating 2 | 5 | 2
  2 - Functioning at high levels, but not at peak - Rating 2 | 5 | 1
  3 - Awake, but relaxed; responsive, but not fully alert - Rating 2 | 0 | 2
  4 - Somewhat foggy, let down - Rating 2 | 0 | 5
  5 - Foggy; losing interest in staying awake; slowed down - Rating 2 | 0 | 0
  6 - Sleepy, woozy, fighting sleep; prefer to lie down - Rating 2 | 0 | 0
  7 - No longer fighting sleep; sleep onset soon - Rating 2 | 0 | 0
  X - Asleep - Rating 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Adverse events were not separated by intervention because no events occurred during the administration of either the experimental or control conditions. All adverse events reported occurred outside of the study visits and were determined to be unrelated to the study interventions. These events were monitored and documented in accordance with protocol guidelines and were not associated with the auditory exposures.
Groups:
- Preferred Music - Visit 1, Nature Sounds - Visit 2; Nature Sounds - Visit 1, Preferred Music - Visit 2: Preferred Music Participants will listen to selected music using over-ear headphones delivered as 10-minute segments at the top of each hour over the course of 3 hours
  Nature Sounds Participants will listen to nature sounds using over-ear headphones delivered as 10-minute segments at the top of each hour over the course of 3 hours
Arm/Group | Preferred Music - Visit 1, Nature Sounds - Visit 2 | Nature Sounds - Visit 1, Preferred Music - Visit 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preferred Music - Visit 1, Nature Sounds - Visit 2 (N=5) | Nature Sounds - Visit 1, Preferred Music - Visit 2 (N=5)
Fall (General disorders) | 2 | 0
Arm Abrasion (General disorders) | 1 | 0
Muscle Strain (General disorders) | 0 | 1
Common cold (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05309369/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05309369/ICF_000.pdf